CLINICAL TRIAL: NCT00499317
Title: Genetic Study of Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS)
Acronym: CP/CPPS
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Catherine Brownstein, Assoc. Professor of Genetics and Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: 04-11-160M; 91208 (Other Grant/Funding Number: Broad Institute)
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Chronic Prostatitis (CP); Chronic Pelvic Pain Syndrome (CPPS); Painful Bladder Syndrome (PBS); Benign Frequency Syndrome (BFS); Interstitial Cystitis
Keywords: Urgency; Frequency; Pelvic pain; Sexual dysfunction; Erectile dysfunction; Painful intercourse
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain; Sexual Dysfunction, Physiological; Erectile Dysfunction; Dyspareunia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample via blood/saliva, bladder tissue and urine samples will be collected and stored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS) is a condition with several causes of which some remain unknown. It is believed that some types of CP may be genetic or passed down (inherited) from one generation to the next.

In this study, we are collecting genetic material and medical information to try to determine if genetic factors play a role in CP/CPPS. We will be collecting DNA (from Blood/Saliva sample) and urine from each participant. Bladder tissue from affected individuals will also be collected. Individuals and families with CP/CPPS will be enrolled. Family members of an individual with CP/CPPS are eligible whether or not they also experience CP/CPPS symptoms.

DETAILED DESCRIPTION:
We would like to determine if chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) has a genetic cause. We will be attempting to further describe the symptoms of CP/CPPS and to correlate them with changes in your genes. We will use several types of genetic testing; linkage analysis, whole exome sequencing and candidate gene studies. Each individual participant will be required to give a DNA sample (via Blood/Saliva), a urine sample and answer questionnaires. Affected participants will also be asked to provide a bladder sample from a clinical biopsy. All samples will be stored. Travel to Boston NOT required.

ELIGIBILITY:
Inclusion Criteria:

* Have symptoms for at least 3 months within the preceding 6 months:
* Pain in the pelvic area
* Urinary frequency and/or
* Urinary urgency and/or
* Sexual dysfunction (erectile dysfunction)
* Have CP/CPPS, Interstitial Cystitis (IC), Bladder Pain Syndrome BPS, or Bladder Fasciculation Syndrome (BFS)
* Be willing to provide a blood/saliva, bladder tissue (from previous biopsy) and urine sample
* Agree to complete several brief questionnaires
* Family member of someone with CP/CPPS, BPS, IC or BFS
* Live in the USA or Canada

Exclusion Criteria:

* Major structural/anatomical urinary tract abnormalities
* Underlying inborn or congenital conditions which affect the urinary tract
* Surgery/chemotherapy in the pelvic area
* Bacterial cause to CP/CPPS or recurrent Urinary tract infections (UTI)
* Traumatic cause to CP/CPPS

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are collecting individuals with a diagnoses of CP/CPPS and their family members (with or without symptoms) from North America (United States and Canada). Preference is given to families with multiple affected individuals (males or females with IC/BPS/CPPS).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Brownstein, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital (BCH), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from individual participants may be shared with other researchers. Other research studies will be approved by our internal review board and participants samples and data will be de-identified.
Supporting Information: SAP, ICF
Time Frame: We will store study information and samples indefinitely and may share this information with future collaborators. All shared samples and data will be de-identified.
Access Criteria: De-identified data may be shared with other CP/CPPS researchers or other BCH researchers

REFERENCES:
- [Background] Propert KJ, Alexander RB, Nickel JC, Kusek JW, Litwin MS, Landis JR, Nyberg LM, Schaeffer AJ; Chronic Prostatitis Collaborative Research Network. Design of a multicenter randomized clinical trial for chronic prostatitis/chronic pelvic pain syndrome. Urology. 2002 Jun;59(6):870-6. doi: 10.1016/s0090-4295(02)01601-1. PMID 12031372
- [Background] Keay SK, Zhang CO. Abnormal Akt signalling in bladder epithelial cell explants from patients with interstitial cystitis/bladder pain syndrome can be induced by antiproliferative factor treatment of normal bladder cells. BJU Int. 2016 Jul;118(1):161-72. doi: 10.1111/bju.13457. Epub 2016 Mar 29. PMID 26919663
- [Result] Dimitrakov JD. A case of familial clustering of interstitial cystitis and chronic pelvic pain syndrome. Urology. 2001 Aug;58(2):281. doi: 10.1016/s0090-4295(01)01138-4. PMID 11489726